CLINICAL TRIAL: NCT05729243
Title: Cytisine: Testing Its Potential as a Therapeutic Strategy for Smoking Cessation Among People With Concurrent Alcohol Use Disorder
Brief Title: Cytisine for Smoking Cessation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 054-2022
Record Dates: First submitted 2023-01-24; First posted 2023-02-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Tobacco Use Disorder; Alcohol Use Disorder; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism; Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytisine (Experimental): Cytisine will be given as 1.5 mg tablet formulations for 25 days.
  The following treatment schedule will be followed:
  * Days 1 to 3: 1.5 mg taken every 2 hours (6 pills (9 mg)/day)
  * Days 4 to 12: 1.5 mg taken every 2.5 hours (5 pills (7.5 mg)/day)
  * Days 13 to 16: 1.5 mg taken every 3 hours (4 pills (6 mg)/day)
  * Days 17 to 20: Taper down to 1 tablet every 5 hours (3 pills (4.5 mg)/day)
  * Days 21 to 25: Taper down to 1-2 tablets daily (1.5-3 mg/day)
  Interventions: Drug: Cytisine
- Placebo (Placebo Comparator): Placebo will be given following the same schedule as the Cytisine Arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cytisine — Cytisine is a nicotinic acetylcholine receptor partial agonist and is a natural health product approved by Health Canada. Cytisine has been used for a long time in Europe for smoking cessation.
  Arms: Cytisine
Other: Placebo — A placebo identical in appearance to cytisine will be used
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of cytisine as a smoking cessation treatment in individuals with concurrent alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years;
* Have TUD assessed by structured clinical interview for DSM-5;
* Have past year AUD (active) assessed by structured clinical interview for DSM-5;
* Report daily cigarette consumption in past month and expired carbon monoxide (CO) measurement ≥10ppm at screening;
* Have Fagerstrom Test of Nicotine Dependence (FTND55) score ≥4;
* Have motivation to quit within 30 days i.e. Contemplation Ladder56 score ≥7;
* Be willing and able to comply with all study procedural and assessment demands;
* Be able to provide voluntary written informed consent.

Exclusion Criteria:

* Report prolonged smoking abstinence in the past month preceding screening;
* Be using other smoking cessation aids
* Enrolled in another smoking cessation program
* Be pregnant, breastfeeding, or intending to become pregnant or breastfeed;
* Exhibit suicidal thoughts or behavior in the past month;
* Enrolled in another study which would interfere with study procedures or represent a potential risk to the participant
* Have a serious unstable psychiatric or medical condition preventing participation in the trial. This includes some forms of schizophrenia, ischemic heart disease, heart failure, arterial hypertension (systolic BP above 150; diastolic BP above 100), cerebrovascular diseases, occlusion of blood vessels, kidney and/or liver disease, hyperthyroidism, ulcer, diabetes, Chromaffin tumours of the adrenal medulla, and gastroesophageal reflux disease (GERD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Frequency and type of adverse events | Total duration of trial (24 weeks)
  To assess the tolerability of cytisine
Rate of retention in the trial: number of sessions completed for each participant and number ofparticipants who withdraw | Total duration of trial (24 weeks)
  To assess the tolerability of cytisine

SECONDARY OUTCOMES:
Point-prevalence abstinence | Week 2 and week 4
  Complete abstinence ("not even a puff") during a designated time period (7 days) prior to assessment. This will be measured at each assessment point (e.g., 2 and 4wk).
Repeated point-prevalence abstinence | Throughout study completion, up to 24 weeks.
  Point-prevalence abstinence at each consecutive assessment point.
Prolonged abstinence | This period will end at the end of treatment (day 25) or at final follow-up.
  Complete abstinence ("not even a puff") after an initial grace period; also known as sustained abstinence.
Prolonged abstinence with lapses | This period will end at the end of treatment (day 25) or at final follow-up.
  Prolonged abstinence after a grace period, but some smoking is allowed (e.g., no more than 5 cigarettes; fewer than seven consecutive days of smoking).
Continuous Abstinence | Throughout study completion, up to 24 weeks.
  Complete abstinence ("not even a puff") beginning on the TQD (i.e., with no grace period) and lasting until the assessment from target quit date (week 2) to end of treatment (day 25) and at final follow up.
Physical dependence to Nicotine in Participants | Throughout study duration (24 weeks)
  The Fagerstrom Test for Nicotine Dependence (FTND) will be used to assess physical dependence in participants.
Nicotine Withdrawal Symptoms in Participants | Throughout study duration (24 weeks)
  The Minnesota Nicotine Withdrawal Scale (MNWS) will be used to assess nicotine withdrawal symptoms.
Nicotine Craving in Participants | Throughout study duration (24 weeks)
  Tiffany Questionnaire of Smoking Urges (QSU) will be used to assess nicotine craving.

OTHER OUTCOMES:
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on anxiety. | Throughout study duration (24 weeks)
  Anxiety will be measured through the General Anxiety Disorder-7 (GAD-7) questionnaire.
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on mood. | Throughout study duration (24 weeks)
  Mood will be measured by the Patient Health Questionnaire-9 (PHQ-9).
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on Quality of Life. | Throughout study duration (24 weeks)
  Quality of Life will be measured through the WHO Disability Assessment Schedule (WHODAS).
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on drinking by collecting the number of drinking days in participants. | Throughout study duration (24 weeks)
  Number of drinking days and drinks per day/drinking day will be collected.
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on drinking by measuring the proportion of heavy drinking days in participants. | Throughout study duration (24 weeks)
  Percent of heavy drinking days (5+/4+ males/females)/very heavy drinking days (10+/8+ males/females) per week and per month will be collected.
Tertiary Endpoints to evaluate the impact of cytisine vs. placebo on drinking by measuring the proportion of participants without heavy drinking days. | Throughout study duration (24 weeks)
  Percent of subjects who are abstinent, percent of subjects with no heavy drinking days and percent of days abstinent will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, Principal Investigator — The Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada